CLINICAL TRIAL: NCT02626104
Title: Bovine Lactoferrin in the Prevention of Antibiotic-associated Diarrhoea in Children - a Randomized Clinical Trial.
Brief Title: Bovine Lactoferrin and Antibiotic-associated Diarrhoea.
Acronym: BLAAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Pharmabest Sp. z o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BLAAD
Record Dates: First submitted 2015-06-29; First posted 2015-12-10 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2015-11

CONDITIONS: Antibiotic Associated Diarrhoea
Keywords: lactoferrin; clostridium difficile; antibiotic associated diarrhoea; children; antibiotic therapy; diarrhoea
MeSH Terms: conditions — Diarrhea | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - Lactoferrin (Experimental): Bovine lactoferrin orally - 100 mg twice a day, for whole antibiotic treatment period.
  Interventions: Dietary Supplement: Bovine lactoferrin
- B - Maltodextrin (Placebo Comparator): Maltodextrin orally - 100 mg twice a day, for whole antibiotic treatment period.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Bovine lactoferrin — The children will be randomly assigned to receive 100 mg of bovine lactoferrin twice a day orally for the whole period of antibiotic therapy.
  Arms: A - Lactoferrin
Dietary Supplement: Maltodextrin — The children will be randomly assigned to receive 100 mg of placebo - maltodextrin twice a day orally for the whole period of antibiotic therapy.
  Arms: B - Maltodextrin

SUMMARY:
This prospective, randomized, parallel-group, double blind, single-center study is to be conducted in the Medical University of Warsaw Public Paediatric Teaching Hospital in following departments: Department of Paediatric Gastroenterology and Nutrition, Department of Paediatrics and Nephrology, Department of Pediatric Pneumonology and Allergy, Department of Pediatrics with Medical Assessment Unit, Admissions Department. It is planned to include a total of 156 children aged between 12 months to 18 years old receiving antibiotic therapy because of acute respiratory tract infection/or urinary tract infection. The children will be randomly assigned to receive 100 mg of bovine lactoferrin or placebo twice a day orally for the whole period of antibiotic therapy. The primary efficacy parameter is occurrence of diarrhea during the antibiotic therapy and two weeks after, defined as > 3 stools a day, a watery or loose stool with/or occurrence of blood in the stool.

ELIGIBILITY:
Inclusion Criteria:

* acute respiratory or urinary infection requiring empiric antibiotic therapy.
* antibiotic treatment started before 24 hours prior to enrollment.
* the consent of parents or legal guardians to participate in the study

Exclusion Criteria:

* severe or generalized bacterial infection
* antibiotic therapy during the last 8 weeks
* use of probiotic during the seven days prior to enrollment
* immune disorders,
* chronic disease of the gastrointestinal tract,
* actual acute or chronic diarrhea,
* intake of iron supplementation,
* cows milk protein allergy
* lack of consent of the parents or legal guardians to participate in the study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Occurence of antibiotic-associated diarrhoea. | Up to 24 days after initiation of antibiotic treatment.
  Occurrence of diarrhea up to 24 days after initiation of antibiotic treatment, defined as > 3 stools a day, a watery or loose stool with/or occurrence of blood in the stool.

SECONDARY OUTCOMES:
Discontinuation of antibiotic treatment due to the antibiotic - diarrhoea. | Up to 10 days after initiation of antibiotic treatment.
Intravenous rehydration due to the antibiotic-associated diarrhea | Up to 24 days after initiation of antibiotic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Albrecht, Ph.D., Study Chair — Department of Paediatric Gastroenterology and Nutrition
Locations (1):
- Medical University of Warsaw's Department of Paediatric Gastroenterology and Nutrition, Warsaw, Masovian Voivodeship, Poland

REFERENCES:
- [Derived] Wronowski MF, Kotowska M, Banasiuk M, Kotowski A, Kuzmicka W, Albrecht P. Bovine Lactoferrin in the Prevention of Antibiotic-Associated Diarrhea in Children: A Randomized Clinical Trial. Front Pediatr. 2021 Jun 7;9:675606. doi: 10.3389/fped.2021.675606. eCollection 2021. PMID 34164360